CLINICAL TRIAL: NCT04704128
Title: Identification de Voies Physiopathologiques et Cibles thérapeutiques Dans la Stomatodynie Primaire (" Burning Mouth Syndrome ") Par la métabolomique Salivaire : étude Cas/témoins
Brief Title: Identification of Pathophysiological Pathways and Therapeutic Targets in Primary Stomatodynia by Salivary Metabolomics
Acronym: SESAME
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI20-SESAME; 2020-A03435-34 (Other: IdRCB); 20.12.14.65838 (Other: SI CNRIPH)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Primary Burning Mouth Syndrome
Keywords: Primary Burning Mouth Syndrome; Salivary metabolomic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: women with primary stomatodynia
  Interventions: Other: Salivic sample
- Control group: women without oral disease
  Interventions: Other: Salivic sample

INTERVENTIONS:
Other: Salivic sample — Collection of total saliva not stimulated

SUMMARY:
Burning mouth syndrome (BMS) is defined by a chronic oral pain affecting especially postmenopausal women. Its physiopathology is still unknown and several hypotheses have been put forward to explain this syndrome, such as neurological, hormonal or inflammatory process. The recent development of salivary metabolomic profiling in oral diseases has led to the identification of potential pathways in such disorders. The aim of this study is to analyze the salivary metabolomic in BMS patients compared to healthy controls.

DETAILED DESCRIPTION:
Burning mouth syndrome (BMS) is defined by a chronic oral pain affecting especially postmenopausal women. Its physiopathology is still unknown and several hypotheses have been put forward to explain this syndrome, such as neurological, hormonal or inflammatory process. The recent development of salivary metabolomic profiling in oral diseases has led to the identification of potential pathways in such disorders. The aim of this study is to analyze the salivary metabolomic in BMS patients compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* For cases : primary Burning Mouth Syndrome, based on the IHS diagnosis criteria
* For cases : being able to realise the salivary collection
* For controls : no primary BMS
* For controls : being able to realise the salivary collection

Exclusion Criteria for both groups:

* Treatment by antibiotics in the previous month
* New treatment in the previous two weeks
* Active smoking
* Active infectious or inflammatory oral disease
* Systemic disease that could have an impact on the salivary metabolome or on the neurological system
* Being under legal guardianship
* Opposition to the processing of personal data

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Regarding the high predominance of this pathology among women and in order to optimize the study homogeneity, only women will be enrolled in this study.
  In the control group, patients will be selected for having close characteristics with cases (pairing for age +/- 5 years and for sex).
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
Comparative analysis of salivary metabolomic profiles between cases (primary BMS) and controls | at inclusion
  metabolites will be measured in saliva by chromatography-mass spectrometry

SECONDARY OUTCOMES:
Comparative analysis of salivary neuropeptides between cases (primary BMS) and controls | at inclusion
  quantitative assessment of levels of neuropeptides (NGF, histamine, tryptase, kallicrein) will be assessed in saliva in cases and controls
Comparative analysis of salivary hormones between cases (primary BMS) and controls | at inclusion
  quantitative assessment of levels of steroid hormones (cortisol, 11-desoxycortisol, DHEA, SDHEA, progesterone, 17-hydroxyprogesterone, testosterone, androstenedione) will be assessed in saliva in cases and controls
Comparative analysis of salivary inflammatory cytokines between cases (primary BMS) and controls | at inclusion
  quantitative assessment of levels of cytokines (IL-2, IL-6, IL-18, TNFα) will be assessed in saliva in cases and controls
Correlation between salivary biomarkers and pain characteristics | at inclusion
  metabolites profile, salivary neuropeptides, hormones and cytokines will be compared according to the category of pain (type I-II-III, neuropathic pain score DN4>4)

CONTACTS AND LOCATIONS:
Overall Officials: Mahtab SAMIMI, MD-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Department of Dermatology, Hospital University of Tours, Tours, France